CLINICAL TRIAL: NCT03807752
Title: The Effect of Supplementation With a Marine Protein Hydrolysate in Patients With Metabolic Syndrome
Brief Title: Marin Protein Hydrolysate and Metabolic Syndrome
Acronym: MPH_MetS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Haukeland University Hospital (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/2163
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Metabolic Syndrome
Keywords: Dietary Supplements; Fish Proteins; Protein Hydrolysates
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: A parallel group randomized, controlled clinical trial for eight weeks
Who Masked: Participant, Care Provider, Investigator
Masking Description: The provider of the dietary supplement deliver the supplement prepared and packed in equal bags (active/placebo) that we hand out to the participants in an randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPH_active (Active Comparator): Daily intake at breakfast of supplementary marine protein hydrolysate (MPH). Random sequence of arms.
  Interventions: Dietary Supplement: MPH_active
- MPH_placebo (Placebo Comparator): Daily intake at breakfast of supplementary placebo. Random sequence of arms.
  Interventions: Dietary Supplement: MPH_placebo

INTERVENTIONS:
Dietary Supplement: MPH_active — One daily intake at breakfast of supplementary marine protein hydrolysate (MPH), a dosage of X mg, duration 8 weeks. The form is powder, flavored with lemon, and to be mixed with 100 ml water. Random sequence of arms.
  Arms: MPH_active
Dietary Supplement: MPH_placebo — One daily intake at breakfast of supplementary placebo, a dosage of X mg, duration 8 weeks. The form is powder, flavored with lemon, and to be mixed with 100 ml water.
  Arms: MPH_placebo

SUMMARY:
Overweight and obesity are increasing global health problems and the most important contributors to morbidity and mortality. The maintenance of long-term weight loss is difficult, and individuals often regain weight after an intervention program is finished. It is of interest to find ways to prevent and alleviate metabolic syndrome (MetS), beyond the known effects of lifestyle modification and weight loss. Fish has been proposed as a food that may have favorable effects on metabolic health. There is evidence that cod, and other marine fish, may contain bioactive peptides that have potentially important health effects in humans. The aim of this study is to investigate the effect of adding a marine protein hydrolysate (MPH) supplement to the diet over an 8-week period in a group of adults with established MetS. The investigators expect that this will lead to beneficial changes in the components of MetS and to an overall healthier metabolic profile.

DETAILED DESCRIPTION:
Overweight and obesity are increasing global health problems and the most important contributors to morbidity and mortality. Obesity (abdominal obesity), together with hyperglycemia, dyslipidemia and hypertension forms a cluster of risk factors that is called the metabolic syndrome (MetS). The first-line therapy for MetS is lifestyle intervention - education on a healthy lifestyle leading to a focus on physical activity and diet, which will improve risk factors closely linked to MetS. The maintenance of long-term weight loss is difficult, and individuals often regain weight after an intervention program stops. It is of interest to find ways to prevent and alleviate MetS, beyond the known effects of lifestyle modification and weight loss. Fish has been proposed as a food that may have favorable effects on metabolic health. Previous intervention studies with fish protein in humans and rodents have shown improved insulin sensitivity and glucose tolerance, reduced cholesterol levels in plasma and reduced blood pressure. Intervention studies investigating the effect of cod have mainly focused on the health effect of consuming the whole fillet. Studies on the remaining part of the fish, the residual material, primarily used for production of animal feed, are scarce. There is evidence that cod, and other marine fish, may contain bioactive peptides that have potentially important health effects in humans. Therefore, it is of interest to investigate the possible effect of a daily supplement of marine protein hydrolysate (MPH), taken over a longer period, in a group of patients with abnormal glucose control. The aim of this study is to investigate the effect of adding a MPH supplement to the diet over an 8-week period in a group of adults with established MetS. The investigators expect that supplementation with MPH will lead to beneficial changes in the components of MetS and an overall healthier metabolic profile.

ELIGIBILITY:
Inclusion Criteria:

Age 40-70 years

* BMI 27-35 kg/m2
* Signed informed consent
* MetS as defined by the presence of at least 3 of the 5 following criteria*:

  * Elevated waist circumference ≥ 94 cm (M), ≥ 80 cm (F)
  * Elevated triglycerides ≥ 1.7 mmol/L (150 mg/dL)
  * Elevated fasting glucose ≥ 5.5 mmol/L (100 mg/dL)
  * Elevated blood pressure S ≥ 130 and/or D ≥85 mmHg
  * Reduced HDL-cholesterol < 1.0 mmol/L (40 mg/dL) (M) <1.3 mmol/L (50 mg/dL) (F)

    * The International Diabetes Foundations (IDF) cut-off points are used.

Exclusion Criteria:

* Suspected allergy against fish or shellfish
* Acute infections (may be reconsidered for inclusion at a later time)
* Chronic disease or therapies that is likely to interfere with the evaluation study results
* Pregnancy, lactation or planning pregnancy during study period
* Substance misuse
* Inability or unwillingness to comply with the requirements of study procedures

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Glucose | At baseline and after 8 weeks, the first sample fasted, thereafter repeated samples every 20 minutes (i.e. -15, 0, 20, 40, 60, 80, 100,120 minutes after baseline).
  Postprandial glucose (mmol/L) change at baseline and after 8 weeks on intervention.

SECONDARY OUTCOMES:
Insulin | At baseline and after 8 weeks, the first sample fasted, thereafter repeated samples every 20 minutes (i.e. -15, 0, 20, 40, 60, 80, 100,120 minutes after baseline).
  Postprandial insulin (mmol/L) change at baseline and after 8 weeks on intervention.
Hormon hunger 1 | At baseline and after 8 weeks, the first sample fasted, thereafter repeated samples (i.e - 15, 0, 20, 40, 80, 120 minutes after baseline).
  Glucagon like peptide 1 (GLP-1) pmol/l at baseline and after 8 weeks on intervention.
Hormon hunger 2 | At baseline and after 8 weeks, the first sample fasted, thereafter repeated samples (i.e - 15, 0, 20, 40, 80, 120 minutes after baseline).
  Ghrelin at baseline and after 8 weeks on intervention.
Body composition 1 | At baseline and after 8 weeks.
  Bioimpedance at baseline and after 8 weeks on intervention.
Body composition 2 | At baseline and after 8 weeks.
  Body mass index at baseline and after 8 weeks on intervention.
Body composition 3 | First at baseline and after 8 weeks.
  Waist circumference at baseline and after 8 weeks on intervention.
Glucose_met | At baseline and after 8 weeks.
  Glycated hemoglobin (HBA1c) at baseline and after 8 weeks on intervention.

OTHER OUTCOMES:
Inflammation | At baseline and after 8 weeks.
  High-sensitive C-reactive protein at baseline and after 8 weeks on intervention.
Hormon 2 | Fasted at baseline and after 8 weeks.
  Adiponectin at baseline and after 8 weeks on intervention.
Hormon 1 | Fasted at baseline and after 8 weeks.
  Leptin at baseline and after 8 weeks on intervention.
Lipid profile 1 | Fasted at baseline and after 8 weeks.
  Triglycerides at baseline and after 8 weeks on intervention.
Lipid profile 2 | Fasted at baseline and after 8 weeks.
  Total cholesterol at baseline and after 8 weeks on intervention.
Lipid profile 3 | Fasted at baseline and after 8 weeks.
  HDL-cholesterol at baseline and after 8 weeks on intervention.
Lipid profile 4 | Fasted at baseline and after 8 weeks.
  LDL-cholesterol at baseline and after 8 weeks on intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne Lihaug Hoff, MD, PhD, Study Director — Helse Møre og Romsdal Hospital Trust
Locations (2):
- Norway (2):
  - Ålesund Hospital, Helse Møre og Romsdal HF, Ålesund
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen C, Dale HF, Hausken T, Hatlebakk JG, Bronstad I, Lied GA, Hoff DAL. The Effect of Supplementation with Low Doses of a Cod Protein Hydrolysate on Satiety Hormones and Inflammatory Biomarkers in Adults with Metabolic Syndrome: A Randomized, Double-Blind Study. Nutrients. 2020 Nov 8;12(11):3421. doi: 10.3390/nu12113421. PMID 33171589
- [Result] Jensen C, Fjeldheim Dale H, Hausken T, Hatlebakk JG, Bronstad I, Lied GA, Hoff DAL. Supplementation with Low Doses of a Cod Protein Hydrolysate on Glucose Regulation and Lipid Metabolism in Adults with Metabolic Syndrome: A Randomized, Double-Blind Study. Nutrients. 2020 Jul 4;12(7):1991. doi: 10.3390/nu12071991. PMID 32635503